CLINICAL TRIAL: NCT06024278
Title: Developing and Pilot Testing Culturally Based Educational Videos for Puerto Rican and African American Home Hospice Caregivers
Brief Title: Developing and Testing Culturally Based Educational Videos for Puerto Rican and African American Home Hospice Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); VNS Health (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-04024661; 3K76AG059997-03S1 (NIH)
Record Dates: First submitted 2023-08-29; First posted 2023-09-06 (Actual); Results first posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-11

CONDITIONS: Caregivers of Patients on Hospice Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- African American Hospice Caregivers (Experimental): Culturally tailored educations videos will be administered to African American participants.
  Interventions: Behavioral: Caregiver educational videos for African American caregivers
- Puerto Rican Hospice Caregivers (Experimental): Culturally tailored educations videos will be administered to Puerto Rican participants.
  Interventions: Behavioral: Caregiver educational videos for Puerto Rican caregivers

INTERVENTIONS:
Behavioral: Caregiver educational videos for African American caregivers — The intervention will be culturally tailored education videos for African American caregivers receiving hospice services.
  Arms: African American Hospice Caregivers
Behavioral: Caregiver educational videos for Puerto Rican caregivers — The intervention will be culturally tailored education videos for Puerto Rican caregivers receiving hospice services.
  Arms: Puerto Rican Hospice Caregivers

SUMMARY:
The investigators hypothesize that culturally based educational videos for Puerto Rican and African American home hospice caregivers will better inform caregivers in managing symptoms, preparedness, self-efficacy, and competence.

DETAILED DESCRIPTION:
The clinical trial for this project is a cross-sectional study conducted with VNS Health hospice, Hospicio Toque de Amor, and Hospicio Luz Celeste. Names of Puerto Rican and African American caregivers receiving home hospice care will be referred to the study team by the site leader/hospice leadership at each hospice. Demographic data will be collected from each caregiver participant. Prior to showing participants the culturally tailored videos, a research member will administer a set of Likert style questions developed by the research team around comfort in managing symptom related issues. The same questions will be administered again post video intervention. In addition, the preparedness scale, chronic pain self-efficacy scale, and caregiving competence scale will be administered to participants pre and post video intervention. The PI will not be involved in the administering the intervention for this study. After the culturally tailored videos have been shown to the participant, a research member will also conduct an open-ended interview about content, reactions, attitudes, usefulness and limitations around each video. Interviews will be conducted in either English and/or Spanish.

ELIGIBILITY:
Inclusion Criteria:

* Family caregivers who identify themselves as Puerto Rican or African American
* English and/or Spanish speaking
* 18 year of age or older
* Currently receiving home hospice services with a patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veerawat Phongtankuel, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (3):
- VNS Health, New York, New York, United States
- Puerto Rico (2):
  - Hospicio Toque De Amor, Manatí, PR
  - Hospicio Luz Celeste, Caguas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (10.47) | 68.1 (12.89) | 61.6 (13.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 10 | 11
  Not Hispanic or Latino | 9 | 0 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 0 | 9
  White | 0 | 4 | 4
  More than one race | 1 | 6 | 7
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Puerto Rico | 0 | 10 | 10
  United States | 10 | 0 | 10
Highest Education Completed [Count of Participants; unit: Participants]
  Graduate Degree | 3 | 1 | 4
  College Degree | 5 | 3 | 8
  Some College | 1 | 2 | 3
  High School or GED | 1 | 2 | 3
  8th grade or less | 0 | 2 | 2
Relationship to Patient [Count of Participants; unit: Participants]
  Spouse/Partner | 1 | 5 | 6
  Child | 7 | 3 | 10
  Relative | 2 | 1 | 3
  Other | 0 | 1 | 1
Religion [Count of Participants; unit: Participants]
  Evangelical | 0 | 4 | 4
  Catholic | 0 | 3 | 3
  Pentecostal | 0 | 1 | 1
  Christian | 4 | 0 | 4
  Protestant | 1 | 0 | 1
  Baptist | 1 | 0 | 1
  Buddhist | 1 | 0 | 1
  Non-denominational | 1 | 0 | 1
  Not religious but spiritual | 1 | 0 | 1
  Not religious nor spiritual | 1 | 2 | 3
Hours per day spent caregiving [Mean (Standard Deviation); unit: hours] | 9.33 (9.05) | 18.9 (6.62) | 14.9 (8.77)
Caregiving Responsibilities - Provided personal care to their care recipient [Count of Participants; unit: Participants] | 9 | 10 | 19
Caregiving Responsibilities - Managed their care recipients' symptoms [Count of Participants; unit: Participants] | 8 | 10 | 18
Caregiving Responsibilities - Managed their care recipients' medications [Count of Participants; unit: Participants] | 8 | 10 | 18
Caregiving Responsibilities - Communicated with hospice providers on their care recipients' behalf [Count of Participants; unit: Participants] | 10 | 10 | 20
Caregiving Responsibilities - Provided emotional support to their care recipient [Count of Participants; unit: Participants] | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Caregivers' Comfort in Managing Shortness of Breath as Assessed by a Likert Scale at Pre-Intervention
Description: Question ranges from 1 (Extremely uncomfortable) to 5 (Very comfortable)
Time Frame: Pre-intervention at Day 1
Population: Per protocol, this measure was analyzed only for the African American hospice caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 10 | 0
score on a scale | 3.0 (1.15) |

2. Primary Outcome: Caregivers' Comfort in Managing Shortness of Breath as Assessed by a Likert Scale at Post-Intervention
Description: Question ranges from 1 (Extremely uncomfortable) to 5 (Very comfortable)
Time Frame: Post-intervention at Day 1
Population: Per protocol, this measure was analyzed only for the African American hospice caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 10 | 0
score on a scale | 4.1 (0.74) |

3. Primary Outcome: Caregivers' Knowledge in Delivering Liquid Medication as Assessed by a Likert Scale at Pre-Intervention
Description: Question ranges from 1 (No knowledge) to 5 (Very knowledgeable)
Time Frame: Pre-intervention at Day 1
Population: Per protocol, this measure was analyzed only for the African American hospice caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 10 | 0
score on a scale | 3.9 (1.37) |

4. Primary Outcome: Caregivers' Knowledge in Delivering Liquid Medication as Assessed by a Likert Scale at Post-Intervention
Description: Question ranges from 1 (No knowledge) to 5 (Very knowledgeable)
Time Frame: Post-intervention at Day 1
Population: Per protocol, this measure was analyzed only for the African American hospice caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 10 | 0
score on a scale | 4.6 (0.52) |

5. Primary Outcome: Caregivers' Knowledge in Caregiver Resources in Hospice as Assessed by a Likert Scale at Pre-Intervention
Description: Question ranges from 1 (No knowledge) to 5 (Very knowledgeable)
Time Frame: Pre-intervention at Day 1
Population: Per protocol, this measure was analyzed only for the African American hospice caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 10 | 0
score on a scale | 3.2 (1.32) |

6. Primary Outcome: Caregivers' Knowledge in Caregiver Resources in Hospice as Assessed by a Likert Scale at Post-Intervention
Description: Question ranges from 1 (No knowledge) to 5 (Very knowledgeable)
Time Frame: Post-intervention at Day 1
Population: Per protocol, this measure was analyzed only for the African American hospice caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 10 | 0
score on a scale | 4.5 (0.53) |

7. Primary Outcome: Caregivers' Comfort in Using Opioids to Treat Pain as Assessed by a Likert Scale at Pre-Intervention
Description: Question ranges from 1 (Extremely uncomfortable) to 5 (Very comfortable)
Time Frame: Pre-intervention at Day 1
Population: Per protocol, this measure was analyzed only for the African American hospice caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 10 | 0
score on a scale | 3.2 (1.81) |

8. Primary Outcome: Caregivers' Comfort in Using Opioids to Treat Pain as Assessed by a Likert Scale at Post-Intervention
Description: Question ranges from 1 (Extremely uncomfortable) to 5 (Very comfortable)
Time Frame: Post-intervention at Day 1
Population: Per protocol, this measure was analyzed only for the African American hospice caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 10 | 0
score on a scale | 4.0 (1.41) |

9. Primary Outcome: Caregivers' Knowledge in Turning a Patient in Bed as Assessed by a Likert Scale at Pre-Intervention
Description: Question ranges from 1 (No knowledge) to 5 (Very knowledgeable)
Time Frame: Pre-intervention at Day 1
Population: Per protocol, this measure was analyzed only for the African American hospice caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 10 | 0
score on a scale | 4.1 (1.66) |

10. Primary Outcome: Caregivers' Knowledge in Turning a Patient in Bed as Assessed by a Likert Scale at Post-Intervention
Description: Question ranges from 1 (No knowledge) to 5 (Very knowledgeable)
Time Frame: Post-intervention at Day 1
Population: Per protocol, this measure was analyzed only for the African American hospice caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 10 | 0
score on a scale | 4.6 (0.70) |

11. Primary Outcome: Caregivers' Knowledge in Recognizing Patients' Agitation and Confusion as Assessed by a Likert Scale at Pre-Intervention
Description: Question ranges from 1 (No knowledge) to 5 (Very knowledgeable)
Time Frame: Pre-intervention at Day 1
Population: Per protocol, this measure was analyzed only for the African American hospice caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 10 | 0
score on a scale | 4.1 (0.88) |

12. Primary Outcome: Caregivers' Knowledge in Recognizing Patients' Agitation and Confusion as Assessed by a Likert Scale at Post-Intervention
Description: Question ranges from 1 (No knowledge) to 5 (Very knowledgeable)
Time Frame: Post-intervention at Day 1
Population: Per protocol, this measure was analyzed only for the African American hospice caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 10 | 0
score on a scale | 4.6 (0.70) |

13. Primary Outcome: Caregivers' Knowledge in Recognizing End-of-life Signs and Symptoms as Assessed by a Likert Scale at Pre-Intervention
Description: Question ranges from 1 (No knowledge) to 5 (Very knowledgeable)
Time Frame: Pre-intervention at Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 10 | 10
score on a scale | 2.9 (1.60) | 3.1 (1.29)

14. Primary Outcome: Caregivers' Knowledge in Recognizing End-of-life Signs and Symptoms as Assessed by a Likert Scale at Post-Intervention
Description: Question ranges from 1 (No knowledge) to 5 (Very knowledgeable)
Time Frame: Post-intervention at Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 10 | 10
score on a scale | 4.4 (0.70) | 3.2 (1.14)

15. Primary Outcome: Caregivers' Comfort in Managing Shortness of Breath Related to Anxiety as Assessed by a Likert Scale at Pre-Intervention
Description: Question ranges from 1 (Extremely uncomfortable) to 5 (Very comfortable)
Time Frame: Pre-intervention at Day 1
Population: Per protocol, this measure was analyzed only for the Puerto Rican hospice caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 0 | 10
score on a scale |  | 3.0 (1.49)

16. Primary Outcome: Caregivers' Comfort in Managing Shortness of Breath Related to Anxiety as Assessed by a Likert Scale at Post-Intervention
Description: Question ranges from 1 (Extremely uncomfortable) to 5 (Very comfortable)
Time Frame: Post-intervention at Day 1
Population: Per protocol, this measure was analyzed only for the Puerto Rican hospice caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 0 | 10
score on a scale |  | 3.5 (1.51)

17. Primary Outcome: Caregivers' Knowledge About Spiritual Resources in Hospice Care as Assessed by a Likert Scale at Pre-Intervention
Description: Question ranges from 1 (No knowledge) to 5 (Very knowledgeable)
Time Frame: Pre-intervention at Day 1
Population: Per protocol, this measure was analyzed only for the Puerto Rican hospice caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 0 | 10
score on a scale |  | 4.4 (0.70)

18. Primary Outcome: Caregivers' Knowledge About Spiritual Resources in Hospice Care as Assessed by a Likert Scale at Post-Intervention
Description: Question ranges from 1 (No knowledge) to 5 (Very knowledgeable)
Time Frame: Post-intervention at Day 1
Population: Per protocol, this measure was analyzed only for the Puerto Rican hospice caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 0 | 10
score on a scale |  | 4.4 (0.84)

19. Primary Outcome: Caregivers' Comfort in Using Opioids Like Morphine to Help Ease Shortness of Breath as Assessed by a Likert Scale at Pre-Intervention
Description: Question ranges from 1 (Extremely uncomfortable) to 5 (Very comfortable)
Time Frame: Pre-intervention at Day 1
Population: Per protocol, this measure was analyzed only for the Puerto Rican hospice caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 0 | 10
score on a scale |  | 3.1 (1.29)

20. Primary Outcome: Caregivers' Comfort in Using Opioids Like Morphine to Help Ease Shortness of Breath as Assessed by a Likert Scale at Post-Intervention
Description: Question ranges from 1 (Extremely uncomfortable) to 5 (Very comfortable)
Time Frame: Post-intervention at Day 1
Population: Per protocol, this measure was analyzed only for the Puerto Rican hospice caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 0 | 10
score on a scale |  | 3.0 (1.70)

21. Primary Outcome: Caregivers' Comfort in Managing Nausea as Assessed by a Likert Scale at Pre-Intervention
Description: Question ranges from 1 (Extremely uncomfortable) to 5 (Very comfortable)
Time Frame: Pre-intervention at Day 1
Population: Per protocol, this measure was analyzed only for the Puerto Rican hospice caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 0 | 10
score on a scale |  | 3.5 (1.58)

22. Primary Outcome: Caregivers' Comfort in Managing Nausea as Assessed by a Likert Scale at Post-Intervention
Description: Question ranges from 1 (Extremely uncomfortable) to 5 (Very comfortable)
Time Frame: Post-intervention at Day 1
Population: Per protocol, this measure was analyzed only for the Puerto Rican hospice caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 0 | 10
score on a scale |  | 3.7 (1.34)

23. Primary Outcome: Caregivers' Comfort in Managing Constipation as Assessed by a Likert Scale at Pre-Intervention
Description: Question ranges from 1 (Extremely uncomfortable) to 5 (Very comfortable)
Time Frame: Pre-intervention at Day 1
Population: Per protocol, this measure was analyzed only for the Puerto Rican hospice caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 0 | 10
score on a scale |  | 4.1 (0.88)

24. Primary Outcome: Caregivers' Comfort in Managing Constipation as Assessed by a Likert Scale at Post-Intervention
Description: Question ranges from 1 (Extremely uncomfortable) to 5 (Very comfortable)
Time Frame: Post-intervention at Day 1
Population: Per protocol, this measure was analyzed only for the Puerto Rican hospice caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 0 | 10
score on a scale |  | 4.2 (0.79)

25. Primary Outcome: Caregivers' Knowledge About Recognizing Caregiver Stress as Assessed by a Likert Scale at Pre-Intervention
Description: Question ranges from 1 (No knowledge) to 5 (Very knowledgeable)
Time Frame: Pre-intervention at Day 1
Population: Per protocol, this measure was analyzed only for the Puerto Rican hospice caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 0 | 10
score on a scale |  | 3.9 (1.10)

26. Primary Outcome: Caregivers' Knowledge About Recognizing Caregiver Stress as Assessed by a Likert Scale at Post-Intervention
Description: Question ranges from 1 (No knowledge) to 5 (Very knowledgeable)
Time Frame: Post-intervention at Day 1
Population: Per protocol, this measure was analyzed only for the Puerto Rican hospice caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 0 | 10
score on a scale |  | 4.0 (0.94)

27. Primary Outcome: Caregivers' Comfort in Coping With Lack of Appetite for Someone at the End of Life as Assessed by a Likert Scale at Pre-Intervention
Description: Question ranges from 1 (Extremely uncomfortable) to 5 (Very comfortable)
Time Frame: Pre-intervention at Day 1
Population: Per protocol, this measure was analyzed only for the Puerto Rican hospice caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 0 | 10
score on a scale |  | 1.7 (1.06)

28. Primary Outcome: Caregivers' Comfort in Coping With Lack of Appetite for Someone at the End of Life as Assessed by a Likert Scale at Post-Intervention
Description: Question ranges from 1 (Extremely uncomfortable) to 5 (Very comfortable)
Time Frame: Post-intervention at Day 1
Population: Per protocol, this measure was analyzed only for the Puerto Rican hospice caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 0 | 10
score on a scale |  | 2.7 (1.49)

29. Primary Outcome: Caregivers' Knowledge in Making Financial Preparations at the End of Life as Assessed by a Likert Scale at Pre-Intervention
Description: Question ranges from 1 (No knowledge) to 5 (Very knowledgeable)
Time Frame: Pre-intervention at Day 1
Population: Per protocol, this measure was analyzed only for the Puerto Rican hospice caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 0 | 10
score on a scale |  | 3.3 (1.57)

30. Primary Outcome: Caregivers' Knowledge in Making Financial Preparations at the End of Life as Assessed by a Likert Scale at Post-Intervention
Description: Question ranges from 1 (No knowledge) to 5 (Very knowledgeable)
Time Frame: Post-intervention at Day 1
Population: Per protocol, this measure was analyzed only for the Puerto Rican hospice caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 0 | 10
score on a scale |  | 4.0 (1.15)

31. Primary Outcome: Caregivers' Comfort in Managing Agitation and Confusion as Assessed by a Likert Scale at Pre-Intervention
Description: Question ranges from 1 (Extremely uncomfortable) to 5 (Very comfortable)
Time Frame: Pre-intervention at Day 1
Population: Per protocol, this measure was analyzed only for the Puerto Rican hospice caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 0 | 10
score on a scale |  | 2.9 (1.45)

32. Primary Outcome: Caregivers' Comfort in Managing Agitation and Confusion as Assessed by a Likert Scale at Post-Intervention
Description: Question ranges from 1 (Extremely uncomfortable) to 5 (Very comfortable)
Time Frame: Post-intervention at Day 1
Population: Per protocol, this measure was analyzed only for the Puerto Rican hospice caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 0 | 10
score on a scale |  | 3.2 (1.40)

33. Secondary Outcome: Caregiver Preparedness Scale Score at Pre-Intervention
Description: An 8-item scale. Each question ranges from 0 (Not at all prepared) to 4 (Very well prepared). Total score can range from 0 to 32 with higher scores are indicative of feeling better prepared for the caregiving role.
Time Frame: Pre-intervention at Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 10 | 10
score on a scale | 23.5 (6.36) | 24.1 (6.19)

34. Secondary Outcome: Caregiver Preparedness Scale Score at Post-Intervention
Description: as for outcome 33
Time Frame: Post-intervention at Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 10 | 10
score on a scale | 28.3 (3.62) | 26.6 (4.01)

35. Secondary Outcome: Caregiving Competence Scale Score at Pre-Intervention
Description: A 4-item scale. Each question ranges from 1 (Not at all competent) to 4 (Very competent)
Time Frame: Pre-intervention at Day 1
Population: Per protocol, this measure was analyzed only for the African American hospice caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 10 | 0
score on a scale | 13.8 (2.15) |

36. Secondary Outcome: Caregiving Competence Scale Score at Post-Intervention
Description: A 4-item scale. Each question ranges from 1 (Not at all competent) to 4 (Very competent)
Time Frame: Post-intervention at Day 1
Population: Per protocol, this measure was analyzed only for the African American hospice caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 10 | 0
score on a scale | 14.3 (2.06) |

37. Secondary Outcome: Chronic Pain Self-Efficacy Scale at Pre-Intervention
Description: A 22-item scale. Each question is rated on a Likert scale between 10 (very uncertain) to 100 (very certain).
Time Frame: Pre-intervention at Day 1
Population: Data was not collected for this measure.
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 0 | 0

38. Secondary Outcome: Chronic Pain Self-Efficacy Scale at Post-Intervention
Description: A 22-item scale. Each question is rated on a Likert scale between 10 (very uncertain) to 100 (very certain).
Time Frame: Post-intervention at Day 1
Population: Data was not collected for this measure.
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 0 | 0

39. Secondary Outcome: Number of Participants Who Provided Qualitative Feedback That Each Video Culturally Tailored for African American Hospice Caregivers Was Helpful at Post-Intervention
Description: Open ended interviews will be conducted to obtain participant feedback around content, attitudes, usefulness and limitations of the videos. Participants will answer questions asking if each video was helpful in improving their knowledge and comfort with managing their care recipient's symptoms.
  Video 1 includes content on managing shortness of breath, delivering liquid medication to a patient, and caregiver resources offered in hospice care. Video 2 includes content on using opioids to treat pain and turning a patient in bed. Video 3 includes content on recognizing agitation and confusion in a patient. Video 4 includes content on recognizing the signs and symptoms when a patient is at the end of life.
Time Frame: Post-intervention at Day 1
Population: 10 African American caregiver participants watched 4 Videos tailored for African American home hospice caregivers and provided qualitative feedback on whether each video was helpful in improving their knowledge and comfort in caregiving.
  Per protocol, this measure was analyzed only for the African American hospice caregivers.
Measure: Count of Participants; unit: Participants
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 10 | 0
Participants
  Video 1 (tailored for African American caregivers) improvement on caregivers' knowledge and comfort | 9 | 0
  Video 2 (tailored for African American caregivers) improvement on caregivers' knowledge and comfort | 9 | 0
  Video 3 (tailored for African American caregivers) improvement on caregivers' knowledge and comfort | 9 | 0
  Video 4 (tailored for African American caregivers) improvement on caregivers' knowledge and comfort | 9 | 0

40. Secondary Outcome: Number of Participants Who Provided Qualitative Feedback That Each Video Culturally Tailored for Puerto Rican Hospice Caregivers Was Helpful at Post-Intervention
Description: Open ended interviews will be conducted to obtain participant feedback around content, attitudes, usefulness and limitations of the videos. Participants will answer questions asking if each video was helpful in improving their knowledge and comfort with managing their care recipient's symptoms.
  Video 1 includes content on managing shortness of breath related to anxiety, using opioids to ease shortness of breath, and spiritual resources offered in hospice care. Video 2 includes content on managing nausea, managing constipation, and recognizing caregiver stress. Video 3 includes content on coping with lack of appetite for someone at the end of life. Video 4 includes content on making financial preparations at the end of life, managing agitation and confusion, and recognizing end-of-life signs and symptoms.
Time Frame: Post-intervention at Day 1
Population: 10 Puerto Rican caregiver participants watched 4 Videos tailored for Puerto Rican home hospice caregivers and provided qualitative feedback on whether each video was helpful in improving their knowledge and comfort in caregiving.
  Per protocol, this measure was analyzed only for the Puerto Rican hospice caregivers.
Measure: Count of Participants; unit: Participants
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
Number analyzed (Participants) | 0 | 10
Participants
  Video 1 (tailored for Puerto Rican caregivers) improvement on caregivers' knowledge and comfort | 0 | 8
  Video 2 (tailored for Puerto Rican caregivers) improvement on caregivers' knowledge and comfort | 0 | 8
  Video 3 (tailored for Puerto Rican caregivers) improvement on caregivers' knowledge and comfort | 0 | 8
  Video 4 (tailored for Puerto Rican caregivers) improvement on caregivers' knowledge and comfort | 0 | 8

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | African American Hospice Caregivers | Puerto Rican Hospice Caregivers
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-17): https://cdn.clinicaltrials.gov/large-docs/78/NCT06024278/Prot_SAP_001.pdf
  • Informed Consent Form (2023-09-19): https://cdn.clinicaltrials.gov/large-docs/78/NCT06024278/ICF_000.pdf